CLINICAL TRIAL: NCT03066804
Title: A 24-week, Randomized, Double-blind, Multi-center, Parallel LCZ696 on NT-proBNP, Exercise Capacity, Symptoms and Safety Compared to Individualized Medical Management of Comorbidities in Patients With Heart Failure and Preserved Ejection Fraction
Brief Title: A Randomized, Double-blind Controlled Study Comparing LCZ696 to Medical Therapy for Comorbidities in HFpEF Patients
Acronym: PARALLAX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLCZ696D2302; 2016-003410-28 (EudraCT Number)
Expanded Access: Available
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Results first posted 2021-02-08 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Cardiovascular Diseases; Heart Failure; Heart failure with Preserved Ejection Fraction; NT-proBNP; 6 MWT; KCCQ; SF-36; NYHA Class; LCZ696; Enalapril; Valsartan; Angiotensin-Converting Enzyme Inhibitors (ACEi); Angiotensin II Type 1 Receptor Blockers (ARB); Renin Angiotensin System Inhibitors (RASi)
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; Enalapril; Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- sacubitril/valsartan (LCZ696) (Experimental): All patients who fulfill the inclusion/exclusion criteria will be stratified before randomization based upon prior therapy for comorbidities to one of 3 strata: ACEi, ARB or no RASi. Patients in the ACEi strata will receive LCZ696 or enalapril. Patients in the ARB strata will receive LCZ696 or valsartan. Patients in the no RASi strata will receive LCZ696 or matching placebo.
  Patients in the ACEi and ARB strata will take two pills twice daily for each dose: one tablet from the LCZ696 pack and one tablet from the comparator pack. Patients in the no RASi strata will take only one tablet twice daily (LCZ696 or matching placebo).
  In the LCZ696 arm, patients will receive active LCZ696 in titrated doses from level 1 up to level 3 (50 mg, 100 mg and 200 mg twice daily orally).
  Interventions: Drug: sacubitril/valsartan; Drug: Placebo to match enalapril; Drug: Placebo to match valsartan
- Comparator (Active Comparator): Patients randomized to the comparator arm will receive either enalapril (ACE stratum) valsartan (ARB stratum) or LCZ696 matching placebo (no RASi stratum).
  Patients in the ACE stratum randomized to comparator, will receive enalapril in titrated doses from level 1 up to level 3 (2.5 mg, 5 mg and 10 mg twice daily).
  Patients in the ARB stratum randomized to comparator will receive valsartan in titrated doses from level 1 up to level 3 (40 mg , 80 mg and 160 mg twice daily).
  Patients in the no RASi stratum randomized to comparator will receive LCZ696 matching placebo.
  Interventions: Drug: Enalapril; Drug: Valsartan; Drug: Placebo to match sacubitril/valsartan

INTERVENTIONS:
Drug: sacubitril/valsartan — Sacubitril/valsartan is available as 24 mg/26 mg, 49 mg/51 mg, 97 mg/103 mg, respectively in tablet form to be taken orally
  Arms: sacubitril/valsartan (LCZ696)
Drug: Enalapril — Enalapril is available as 2.5 mg, 5 mg, and 10 mg tablet form to be taken orally
  Arms: Comparator
Drug: Valsartan — Valsartan is available as 40 mg, 80 mg, 160 mg tablet form to be taken orally
  Arms: Comparator
Drug: Placebo to match sacubitril/valsartan — Placebo to match LCZ696 50 mg, 100 mg, 200 mg tablet form to be taken orally
  Arms: Comparator
Drug: Placebo to match enalapril — Placebo to match enalapril 2.5 mg, 5 mg, 10 mg tablet form to be taken orally
  Arms: sacubitril/valsartan (LCZ696)
Drug: Placebo to match valsartan — Placebo to match valsartan 40 mg, 80 mg, 160 mg tablet form to be taken orally
  Arms: sacubitril/valsartan (LCZ696)

SUMMARY:
The purpose of this study is to demonstrate the superiority of LCZ696 over individualized medical therapy for comorbidities in reducing N-terminal pro-brain natriuretic peptide (NT-proBNP) and improving exercise capacity and HF symptoms in patients with heart failure with preserved ejection fraction (HFpEF).

DETAILED DESCRIPTION:
This study was a 24-week, randomized, double-blind, multi-center, parallel group, active controlled study to evaluate sacubitril/valsartan compared to individualized medical therapy on NT proBNP, exercise capacity, symptoms and QoL in patients with heart failure and preserved left ventricular ejection (HFpEF) fraction (LVEF > 40%). Patients were initially stratified into one of three strata according to prior treatment for comorbidities: Angiotensin converting enzyme inhibitor (ACEi), angiotensin receptor blocker (ARB) or no prior renin angiotensin system inhibitors (RASi). Patients in each stratum were randomized in a 1:1 ratio and received either sacubitril/valsartan or comparator (i.e.

enalapril for patients in ACEi strata, valsartan for patients in the ARB strata and placebo for patients in the No RASi strata). There was no designated proportion of patients planned in each stratum; the strata were populated based upon the patient's prior treatment regimen. The study consisted of a screening epoch of up to 2 weeks and a randomized treatment epoch of 24 weeks, which included a 1 to 4 week study drug up-titration epoch followed by a 20 to 23 week maintenance epoch. Uptitration to target doses was recommended to occur within the first four weeks of the study, and was performed by Investigator's discretion based on the patient's clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular ejection fraction (LVEF) >40% by echo within 6 months prior to study entry or during the screening epoch
* Symptom(s) of heart failure (HF) requiring treatment with diuretics (including loop, or thiazide diuretics, or mineralocorticoid antagonist [MRAs]) for at least 30 days prior to study entry
* NYHA class II-IV
* Structural heart disease (left atrial enlargement or left ventricular hypertrophy) documented by echocardiogram.
* NT-proBNP > 220 pg/mL for patients with no atrial fibrillation/atrial flutter (AF) or >600 pg/mL for patients with AF
* KCCQ clinical summary score < 75
* Patients on ACEi or ARB therapy must have a history of HTN

Exclusion Criteria:

* Any prior measurement of LVEF ≤ 40%, under stable conditions
* Acute coronary syndrome (including MI), cardiac surgery, other major CV surgery within 3 months , or urgent percutaneous coronary intervention (PCI) within 3 months or an elective PCI within 30 days prior to study entry
* Any clinical event within the 6 months prior to Visit 1 that could have reduced the LVEF (eg MI, coronary artery bypass graft [CABG]), unless an echo measurement was performed after the event confirming the LVEF to be >40%
* Current (within 30 days from Visit 1) acute decompensated HF requiring therapy.
* Current (within 30 days from Visit 1) use of renin inhibitor(s), dual RAS blockade or LCZ696
* History of hypersensitivity to LCZ696 or its components
* Patients with a known history of angioedema
* Walk distance primarily limited by non-cardiac comorbid conditions at study entry
* Alternative reason for shortness of breath such as: significant pulmonary disease or severe COPD, hemoglobin (Hgb) <10 g/dL males and < 9.5 g/dL females, or body mass index (BMI) > 40 kg/m^2.
* Systolic blood pressure (SBP) ≥ 180 mmHg at study entry, or SBP >150 mmHg and <180 mmHg at study entry unless the patient is receiving 3 or more antihypertensive drugs, or SBP < 110 mmHg at study entry.
* Patients with HbA1c > 7.5% not treated for diabetes
* Patients with prior major organ transplant or intent to transplant (ie on transplant list)
* eGFR < 30 ml/min/1.73 m^2 as measured by MDRD at screening
* Serum potassium > 5.2 mmol /L (or equivalent plasma potassium value) at study entry
* History or presence of any other disease with a life expectancy of < 3 years
* Pregnant or nursing women or women of child-bearing potential unless they are using highly effective methods of contraception

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2572 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (321):
- United States (32):
  - Novartis Investigative Site, Andalusia, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Santa Ana, California
  - Novartis Investigative Site, Sylmar, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Stamford, Connecticut
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Thomasville, Georgia
  - Novartis Investigative Site, Arlington Heights, Illinois
  - Novartis Investigative Site, Alexandria, Louisiana
  - Novartis Investigative Site, Chalmette, Louisiana
  - Novartis Investigative Site, Houma, Louisiana
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Corvallis, Oregon
  - Novartis Investigative Site, Abington, Pennsylvania
  - Novartis Investigative Site, Sioux Falls, South Dakota
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Lufkin, Texas
  - Novartis Investigative Site, Tomball, Texas
  - Novartis Investigative Site, Falls Church, Virginia
  - Novartis Investigative Site, Seattle, Washington
- Argentina (12):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, Posadas, Misiones Province
  - Novartis Investigative Site, Salta, Salta Province
  - Novartis Investigative Site, San Miguel de Tucumán, San Miguel de Tucuman
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Formosa
  - Novartis Investigative Site, San Luis
  - Novartis Investigative Site, Santa Fe
- Austria (5):
  - Novartis Investigative Site, Braunau am Inn
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Hall in Tirol
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
- Belgium (5):
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Heusden-Zolder
  - Novartis Investigative Site, Huy
  - Novartis Investigative Site, Kortrijk
- Brazil (10):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Canoas, Rio Grande do Sul
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Blumenau, Santa Catarina
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São José do Rio Preto, São Paulo
- Bulgaria (8):
  - Novartis Investigative Site, Burgas
  - Novartis Investigative Site, Pazardzhik
  - Novartis Investigative Site, Pernik
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Shumen
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Veliko Tarnovo
- Canada (5):
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Oakville, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, St-Georges Beauce, Quebec
- Colombia (5):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Cali, Valle del Cauca Department
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Montería
  - Novartis Investigative Site, San Gil
- Czechia (18):
  - Novartis Investigative Site, Brandýs nad Labem, Czech Republic
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Český Krumlov, Czech Republic
  - Novartis Investigative Site, Jablonec nad Nisou, Czech Republic
  - Novartis Investigative Site, Kroměříž, Czech Republic
  - Novartis Investigative Site, Liberec, Czech Republic
  - Novartis Investigative Site, Louny, Czech Republic
  - Novartis Investigative Site, Pardubice, Czech Republic
  - Novartis Investigative Site, Pilsen, Czech Republic
  - Novartis Investigative Site, Svitavy, Czech Republic
  - Novartis Investigative Site, Tábor, Czech Republic
  - Novartis Investigative Site, Třebíč, Czech Republic
  - Novartis Investigative Site, Jihlava, CZE
  - Novartis Investigative Site, Policska, CZE
  - Novartis Investigative Site, Kolín
  - Novartis Investigative Site, Olomouc Lazce
  - Novartis Investigative Site, Přerov
  - Novartis Investigative Site, Valašské Meziříčí
- Denmark (3):
  - Novartis Investigative Site, Copenhagen NV
  - Novartis Investigative Site, Hvidovre
  - Novartis Investigative Site, Randers
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- France (10):
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Corbeil-Essonnes
  - Novartis Investigative Site, Le Coudray
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Tourcoing
  - Novartis Investigative Site, Valenciennes
- Germany (56):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Essen, DEU
  - Novartis Investigative Site, Detmold, North Rhine-Westphalia
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Bad Homburg
  - Novartis Investigative Site, Bad Oeynhausen
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Brüel
  - Novartis Investigative Site, Buch
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Coburg
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Elsterwerda
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Fürth
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Haßloch
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Koeln-Nippes
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Lüneburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Munich
  - Novartis Investigative Site, Mühldorf
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neuruppin
  - Novartis Investigative Site, Nienburg
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Papenburg
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Riesa
  - Novartis Investigative Site, Rodgau
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rotenburg an der Fulda
  - Novartis Investigative Site, Rüsselsheim am Main
  - Novartis Investigative Site, Schwäbisch Hall
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Stadtlohn
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wallerfing
  - Novartis Investigative Site, Wattenscheid
  - Novartis Investigative Site, Wedel
  - Novartis Investigative Site, Wismar
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (4):
  - Novartis Investigative Site, Budapest, HUN
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Mosanmagyarovar
  - Novartis Investigative Site, Szeged
- India (9):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, Manipal, Karnataka
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Bikaner, Rajasthan
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, India
- Israel (6):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Hadera
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
- Italy (11):
  - Novartis Investigative Site, Cortona, AR
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Legnano, MI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Sesto San Giovanni, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Rovigo, RO
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Cona
  - Novartis Investigative Site, San Vito al Tagliamento
- Latvia (4):
  - Novartis Investigative Site, Liepāja, LVA
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Ogre
  - Novartis Investigative Site, Riga
- Lithuania (3):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Vilnius
- Mexico (3):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Querétaro
  - Novartis Investigative Site, San Luis Potosí City
- Netherlands (11):
  - Novartis Investigative Site, Almelo
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Deventer
  - Novartis Investigative Site, Doetinchem
  - Novartis Investigative Site, Gouda
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Hardenberg
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Stadskanaal
  - Novartis Investigative Site, Tilburg
  - Novartis Investigative Site, Venlo
- Peru (7):
  - Novartis Investigative Site, Trujillo, La Libertad
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, Lima Cercado, Lima region
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, San Miguel, Lima region
  - Novartis Investigative Site, Callao
- Portugal (6):
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Penafiel
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Viana do Castelo
  - Novartis Investigative Site, Vila Real
- Romania (10):
  - Novartis Investigative Site, Bucharest, District 4
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Bacau
  - Novartis Investigative Site, Baia Mare
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Craiova
  - Novartis Investigative Site, Piteşti
  - Novartis Investigative Site, Târgovişte
  - Novartis Investigative Site, Târgu Mureş
  - Novartis Investigative Site, Timișoara
- Russia (11):
  - Novartis Investigative Site, Gatchina
  - Novartis Investigative Site, Ivanovo
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Perm
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Tyumen
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Serbia (5):
  - Novartis Investigative Site, Belgrade
  - Novartis Investigative Site, Kamenitz
  - Novartis Investigative Site, Kragujevac
  - Novartis Investigative Site, Niš
  - Novartis Investigative Site, Niška Banja
- Slovakia (17):
  - Novartis Investigative Site, Námestovo, Slovak Republic
  - Novartis Investigative Site, Prešov, Slovak Republic
  - Novartis Investigative Site, Bratislava, SVK
  - Novartis Investigative Site, Handlová, SVK
  - Novartis Investigative Site, Bardejov
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Dolný Kubín
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Lučenec
  - Novartis Investigative Site, Moldava nad Bodvou
  - Novartis Investigative Site, Nitra
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Považská Bystrica
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Snina
  - Novartis Investigative Site, Svidník
  - Novartis Investigative Site, Trnava
- Spain (17):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Huelva, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Puerto Real, Cadiz
  - Novartis Investigative Site, Villamartín, Cadiz
  - Novartis Investigative Site, Lleida, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, San Sebastián de los Reyes, Madrid
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Manises, Valencia
  - Novartis Investigative Site, Torrevieja (Alicante), Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Las Palmas de Gran Canarias
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Thailand (4):
  - Novartis Investigative Site, Muang, Muang
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Ubon Ratchathani
- Turkey (Türkiye) (12):
  - Novartis Investigative Site, Eskişehir, Meselik
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Aydin
  - Novartis Investigative Site, Bursa
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Sivas
  - Novartis Investigative Site, Talas / Kayseri
- United Kingdom (9):
  - Novartis Investigative Site, High Wycombe, Buckinghamshire
  - Novartis Investigative Site, Stockton-on-Tees, Cleveland
  - Novartis Investigative Site, Chesterfield, Derbyshire
  - Novartis Investigative Site, Craigavon, Northern Ireland
  - Novartis Investigative Site, Wansford, Peterborough
  - Novartis Investigative Site, Addlestone, Surrey
  - Novartis Investigative Site, Sunderland, Tyne and Wear
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, York

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Pieske B, Wachter R, Shah SJ, Baldridge A, Szeczoedy P, Ibram G, Shi V, Zhao Z, Cowie MR; PARALLAX Investigators and Committee members. Effect of Sacubitril/Valsartan vs Standard Medical Therapies on Plasma NT-proBNP Concentration and Submaximal Exercise Capacity in Patients With Heart Failure and Preserved Ejection Fraction: The PARALLAX Randomized Clinical Trial. JAMA. 2021 Nov 16;326(19):1919-1929. doi: 10.1001/jama.2021.18463. PMID 34783839
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=740

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2572 participants were randomized in a 1:1 ratio to receive either sacubitril/valsartan or Individualized Medical Therapy (IMT).
Pre-assignment Details: A total of 2572 participants were randomized in a 1:1 ratio to receive either sacubitril/valsartan or Individualized Medical Therapy (IMT).
Groups:
- Sacubitril/Valsartan (LCZ696): All patients who fulfilled the inclusion/exclusion criteria were stratified before randomization based upon prior therapy for comorbidities to one of 3 strata: ACEi, ARB or no RASi.
- Individualized Medical Therapy (IMT) Comparator: Patients randomized to the comparator arm received either enalapril (ACE stratum) valsartan (ARB stratum) or LCZ696 matching placebo (no RASi stratum).
Period: Overall Study
Arm/Group | Sacubitril/Valsartan (LCZ696) | Individualized Medical Therapy (IMT) Comparator
Started | 1286 | 1286
Completed | 1235 | 1236
Not Completed | 51 | 50
Not completed — Physician Decision | 0 | 4
Not completed — Death | 23 | 17
Not completed — Withdrawal by Subject | 19 | 25
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 2 | 3
Not completed — Technical problems | 5 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set was the primary efficacy population used in the analyses for all efficacy endpoints and included all randomized patients except 6 patients (5 in sacubitril/valsartan group and 1 in IMT group) excluded due to misrandomization or misstratification.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sacubitril/Valsartan (LCZ696) | Individualized Medical Therapy (IMT) Comparator | Total
Number analyzed (Participants) | 1281 | 1285 | 2566
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 196 | 221 | 417
  >=65 years | 1085 | 1064 | 2149
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 643 | 658 | 1301
  Male | 638 | 627 | 1265
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 1112 | 1117 | 2229
  Black | 11 | 16 | 27
  Asian | 56 | 59 | 115
  Native American | 39 | 33 | 72
  Pacific Islander | 0 | 1 | 1
  Unknown | 4 | 3 | 7
  Other | 59 | 56 | 115

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) at Week 12
Description: To demonstrate that LCZ696 is superior to individualized medical therapy for comorbidities in reducing NT-proBNP from baseline at Week 12 in patients with HFpEF
Time Frame: Baseline, week 12
Population: Full Analysis Set: This outcome measure represents patients with non-missing change from baseline in log transformed NT-proBNP at Week 12. The model was fitting using change from baseline in log transformed NT-proBNP, and produced a difference in mean change from baseline in log transformed NT-proBNP, which was then transformed back to geometric mean ratio to baseline using an exponential transformation.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Sacubitril/Valsartan (LCZ696) | Individualized Medical Therapy (IMT) Comparator
Number analyzed (Participants) | 1203 | 1216
Ratio | 0.8218 [0.7955 to 0.8489] | 0.9828 [0.9515 to 1.0151]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (LCZ696) vs Individualized Medical Therapy (IMT) Comparator; Week 12; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Geometric Mean Ratio = 0.8362, 95% CI 2-sided [0.7987 to 0.8754]

2. Primary Outcome: Change From Baseline in 6 Minute Walk Distance (6MWD) at Week 24
Description: Change from baseline in 6-minute walk distance (6MWD) will be reported at Week 24. The 6 MWT will be performed in accordance with the guidelines of the American Thoracic Society 2002.
Time Frame: Baseline, week 24
Population: Subset of Full Analysis Set: This outcome measure was analyzed on patients with a Baseline 6MWD from 100 meters to 450 meters.
Measure: Mean (95% Confidence Interval); unit: Meters
Arm/Group | Sacubitril/Valsartan (LCZ696) | Individualized Medical Therapy (IMT) Comparator
Number analyzed (Participants) | 1082 | 1075
Meters | 9.6935 [5.4310 to 13.9559] | 12.1920 [7.9202 to 16.4638]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (LCZ696) vs Individualized Medical Therapy (IMT) Comparator; Test type: Superiority; p = 0.4164, Mixed Models Analysis; Mean Difference (Net) = -2.4985, 95% CI 2-sided [-8.5267 to 3.52297]

3. Secondary Outcome: Mean Change From Baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) Clinical Summary Score (CSS) at Week 24
Description: The KCCQ is a self-administered questionnaire that requires 4 to 6 minutes to complete. It contains 23 items, covering physical function, clinical symptoms, social function, self-efficacy and knowledge, and Quality of Life (QoL). The CSS is a combined score based upon the clinical symptoms and physical function domains of the questionnaire. Scores are transformed to a range of 0 - 100, in which higher scores reflect better health status.
Time Frame: Baseline, Week 24
Population: Full Analysis Set: This outcome measure represents patients with both baseline KCCQ Clinical Symptom Scores (CSS) and Week 24 KCCQ CSS observed and non-missing covariates.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Sacubitril/Valsartan (LCZ696) | Individualized Medical Therapy (IMT) Comparator
Number analyzed (Participants) | 1207 | 1210
Scores on a scale | 12.3399 [11.3151 to 13.3647] | 11.8168 [10.7922 to 12.8415]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (LCZ696) vs Individualized Medical Therapy (IMT) Comparator; Test type: Superiority; p = 0.4791, Mixed Models Analysis; Mean Difference (Net) = 0.5231, 95% CI 2-sided [-0.9258 to 1.9720]

4. Secondary Outcome: Percentage of Patients With ≥ 5-points Deterioration in KCCQ Clinical Symptom Score(CSS) at Week 24
Description: Percentage of patients with KCCQ CSS deterioration ≥ 5-points will be reported at Week 24. The KCCQ is a self-administered questionnaire that requires 4 to 6 minutes to complete. It contains 23 items, covering physical function, clinical symptoms, social function, self-efficacy and knowledge, and Quality of Life (QoL). The CSS is a combined score based upon the clinical symptoms and physical function domains of the questionnaire. Scores are transformed to a range of 0 - 100, in which higher scores reflect better health status.
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Sacubitril/Valsartan (LCZ696) | Individualized Medical Therapy (IMT) Comparator
Number analyzed (Participants) | 1207 | 1210
Percentage of participants | 15.49 | 16.69
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (LCZ696) vs Individualized Medical Therapy (IMT) Comparator; Test type: Superiority; p = 0.5294, longitudinal binary logistic regression; Odds Ratio (OR) = 0.8993, 95% CI 2-sided [0.6461 to 1.2518]

5. Secondary Outcome: Percentage of Patients With ≥ 5-points Improvement in KCCQ Clinical Symptom Score(CSS) at Week 24
Description: Percentage of patients with KCCQ CSS improvement ≥ 5-points will be reported at Week 24. The KCCQ is a self-administered questionnaire that requires 4 to 6 minutes to complete. It contains 23 items, covering physical function, clinical symptoms, social function, self-efficacy and knowledge, and Quality of Life (QoL). The CSS is a combined score based upon the clinical symptoms and physical function domains of the questionnaire. Scores are transformed to a range of 0 - 100, in which higher scores reflect better health status.
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Sacubitril/Valsartan (LCZ696) | Individualized Medical Therapy (IMT) Comparator
Number analyzed (Participants) | 1207 | 1210
Percentage of participants | 67.94 | 65.70
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (LCZ696) vs Individualized Medical Therapy (IMT) Comparator; Test type: Superiority; p = 0.4938, longitudinal binary logistic regression; Odds Ratio (OR) = 1.1060, 95% CI 2-sided [0.8287 to 1.4760]

6. Secondary Outcome: Change From Baseline in NYHA Functional Class at Week 24
Description: NYHA classification is a subjective physician's assessment of patient's functional capacity and symptomatic status and can change frequently over time.
  Class I - No limitation of physical activity. Ordinary physical activity does not cause symptoms of HF Class II - Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in symptoms of HF Class III - Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes symptoms of HF Class IV - Unable to carry on any physical activity without symptoms of HF, or symptoms of HF at rest
  The NYHA class change will be analyzed as a three category ordinal variable with levels: "improved", "unchanged", and "worsened", defined by at least one class improvement, no change, at least one class worsening, in NYHA class, respectively.
Time Frame: Baseline, week 24
Population: Full Analysis Set: This outcome measure represents patients with both a baseline NYHA class and NYHA class at the visit observed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sacubitril/Valsartan (LCZ696) | Individualized Medical Therapy (IMT) Comparator
Number analyzed (Participants) | 1228 | 1229
Percentage of Participants
  Improved | 23.62 | 24.00
  Unchanged | 72.23 | 71.68
  Worsened | 4.15 | 4.31
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (LCZ696) vs Individualized Medical Therapy (IMT) Comparator; Test type: Superiority; p = 0.8314, Proportional cumulative odds model; Odds Ratio (OR) = 0.9798, 95% CI 2-sided [0.8122 to 1.1820]

7. Secondary Outcome: Change From Baseline in The Short Form 36 Health Survey (SF-36) Physical Component Summary (PCS) Score at Week 24
Description: The SF-36 PCS score reflects the measure of quality of life based on the 36 questions which evaluate the person's physical, emotional, and mental status, including general health. Specifically, the SF-36 PCS score focuses on assessing the person's physical status. The score ranges from 0 to 100 with a higher score indicating a better status of physical wellbeing (range = 0 "worst"-100 "best").
Time Frame: Baseline, Week 24
Population: Full Analysis Set: This outcome measure represents patients with non-missing change from baseline in SF-36 PCS at Week 24.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Sacubitril/Valsartan (LCZ696) | Individualized Medical Therapy (IMT) Comparator
Number analyzed (Participants) | 1185 | 1191
Scores on a scale | 2.5405 [2.0787 to 3.0023] | 2.6975 [2.2360 to 3.1590]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (LCZ696) vs Individualized Medical Therapy (IMT) Comparator; Test type: Superiority; p = 0.6370, Mixed Models Analysis; Mean Difference (Net) = -0.1570, 95% CI [-0.8093 to 0.4953]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of approx. 2 years.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment. AEs were collected and analyzed based on the treatment arm (LCZ696 vs IMT) which the patient was randomized to, regardless of dose level. Hence no dose-specific analysis were performed. Eight patients were excluded from enrolled set [2572], as they did not receive any study treatment (6 patients in the LCZ696 arm and 2 patients in the IMT arm).
Groups:
- Individualized Medical Therapy (IMT): Patients randomized to the comparator arm received either enalapril (ACE stratum) valsartan (ARB stratum) or LCZ696 matching placebo (no RASi stratum).
- Total: Total
Arm/Group | Sacubitril/Valsartan (LCZ696) | Individualized Medical Therapy (IMT) | Total
All-Cause Mortality (participants affected / at risk) | 23/1280 | 17/1284 | 40/2564
Serious Adverse Events (participants affected / at risk) | 186/1280 | 191/1284 | 377/2564
Other Adverse Events (participants affected / at risk) | 964/1280 | 832/1284 | 1796/2564
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sacubitril/Valsartan (LCZ696) (N=1280) | Individualized Medical Therapy (IMT) (N=1284) | Total (N=2564)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 4 | 1 | 5
Acute myocardial infarction (Cardiac disorders) | 2 | 4 | 6
Angina pectoris (Cardiac disorders) | 8 | 8 | 16
Angina unstable (Cardiac disorders) | 6 | 7 | 13
Aortic valve disease (Cardiac disorders) | 0 | 1 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 13 | 17 | 30
Atrial flutter (Cardiac disorders) | 4 | 2 | 6
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 2 | 3 | 5
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 2 | 3
Cardiac arrest (Cardiac disorders) | 1 | 1 | 2
Cardiac failure (Cardiac disorders) | 21 | 31 | 52
Cardiac failure acute (Cardiac disorders) | 3 | 9 | 12
Cardiac failure chronic (Cardiac disorders) | 2 | 1 | 3
Cardiac failure congestive (Cardiac disorders) | 2 | 7 | 9
Cardiac perforation (Cardiac disorders) | 0 | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 1
Cor pulmonale acute (Cardiac disorders) | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 4 | 1 | 5
Dressler's syndrome (Cardiac disorders) | 1 | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 1 | 2
Mitral valve incompetence (Cardiac disorders) | 1 | 1 | 2
Myocardial infarction (Cardiac disorders) | 1 | 4 | 5
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 2
Pericardial effusion (Cardiac disorders) | 1 | 0 | 1
Sinus arrest (Cardiac disorders) | 1 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Mitochondrial myopathy (Congenital, familial and genetic disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 1
Vestibular ataxia (Ear and labyrinth disorders) | 0 | 1 | 1
Cataract (Eye disorders) | 1 | 2 | 3
Eye haemorrhage (Eye disorders) | 1 | 0 | 1
Iris neovascularisation (Eye disorders) | 1 | 0 | 1
Macular hole (Eye disorders) | 0 | 1 | 1
Retinal artery occlusion (Eye disorders) | 0 | 1 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 2 | 1 | 3
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 1 | 2
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 2
Cardiac death (General disorders) | 2 | 0 | 2
Chest pain (General disorders) | 1 | 1 | 2
Death (General disorders) | 0 | 2 | 2
Fatigue (General disorders) | 0 | 1 | 1
Gait disturbance (General disorders) | 1 | 0 | 1
Generalised oedema (General disorders) | 0 | 1 | 1
Malaise (General disorders) | 0 | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2 | 2
Oedema peripheral (General disorders) | 1 | 2 | 3
Pyrexia (General disorders) | 0 | 1 | 1
Sudden death (General disorders) | 0 | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 1 | 2
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 3
Hepatic congestion (Hepatobiliary disorders) | 0 | 1 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 2 | 5
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 3 | 0 | 3
Cholangitis infective (Infections and infestations) | 0 | 1 | 1
Cutaneous leishmaniasis (Infections and infestations) | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 1 | 1
Dengue fever (Infections and infestations) | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1 | 1
Erysipelas (Infections and infestations) | 2 | 3 | 5
Gastroenteritis (Infections and infestations) | 2 | 1 | 3
Hepatitis C (Infections and infestations) | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 1 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 1
Localised infection (Infections and infestations) | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 0 | 3
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 13 | 13 | 26
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 1
Post procedural sepsis (Infections and infestations) | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Sepsis (Infections and infestations) | 2 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 1 | 5
Wound infection (Infections and infestations) | 0 | 1 | 1
Agitation postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 4 | 4
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fractured ischium (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 2 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 1 | 2
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 2 | 3
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Blood urine present (Investigations) | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Carotid artery aneurysm (Nervous system disorders) | 0 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 2
Dementia (Nervous system disorders) | 0 | 1 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 1
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 1 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 6 | 6
Parkinson's disease (Nervous system disorders) | 0 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 2 | 2 | 4
Transient ischaemic attack (Nervous system disorders) | 4 | 0 | 4
Device breakage (Product Issues) | 1 | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 7 | 11
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Nephritic syndrome (Renal and urinary disorders) | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 0 | 3
Renal impairment (Renal and urinary disorders) | 2 | 0 | 2
Renal injury (Renal and urinary disorders) | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 2 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 7
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Accelerated hypertension (Vascular disorders) | 1 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1 | 1
Aortic stenosis (Vascular disorders) | 1 | 1 | 2
Arterial rupture (Vascular disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Haematoma (Vascular disorders) | 1 | 2 | 3
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 2 | 1 | 3
Hypertensive urgency (Vascular disorders) | 0 | 2 | 2
Hypotension (Vascular disorders) | 6 | 2 | 8
Iliac artery stenosis (Vascular disorders) | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1
Peripheral artery occlusion (Vascular disorders) | 1 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 1
Shock (Vascular disorders) | 1 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1 | 1
Thrombosis (Vascular disorders) | 1 | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sacubitril/Valsartan (LCZ696) (N=1280) | Individualized Medical Therapy (IMT) (N=1284) | Total (N=2564)
Anaemia (Blood and lymphatic system disorders) | 17 | 28 | 45
Atrial fibrillation (Cardiac disorders) | 44 | 43 | 87
Cardiac failure (Cardiac disorders) | 34 | 43 | 77
Diarrhoea (Gastrointestinal disorders) | 43 | 42 | 85
Fatigue (General disorders) | 38 | 21 | 59
Oedema peripheral (General disorders) | 43 | 35 | 78
Bronchitis (Infections and infestations) | 29 | 35 | 64
Influenza (Infections and infestations) | 33 | 23 | 56
Nasopharyngitis (Infections and infestations) | 35 | 60 | 95
Urinary tract infection (Infections and infestations) | 49 | 35 | 84
Blood creatinine increased (Investigations) | 27 | 22 | 49
Blood potassium increased (Investigations) | 26 | 10 | 36
Glomerular filtration rate decreased (Investigations) | 137 | 150 | 287
Urine albumin/creatinine ratio increased (Investigations) | 157 | 97 | 254
Urine protein/creatinine ratio increased (Investigations) | 66 | 65 | 131
Hyperkalaemia (Metabolism and nutrition disorders) | 148 | 138 | 286
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 | 21 | 56
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 26 | 53
Dizziness (Nervous system disorders) | 70 | 63 | 133
Headache (Nervous system disorders) | 18 | 30 | 48
Haematuria (Renal and urinary disorders) | 145 | 104 | 249
Microalbuminuria (Renal and urinary disorders) | 26 | 19 | 45
Proteinuria (Renal and urinary disorders) | 121 | 84 | 205
Renal failure (Renal and urinary disorders) | 49 | 38 | 87
Renal impairment (Renal and urinary disorders) | 148 | 110 | 258
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 25 | 66
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 47 | 46 | 93
Pruritus (Skin and subcutaneous tissue disorders) | 27 | 10 | 37
Hypertension (Vascular disorders) | 42 | 81 | 123
Hypotension (Vascular disorders) | 176 | 69 | 245

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT03066804/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT03066804/SAP_001.pdf